CLINICAL TRIAL: NCT05841563
Title: Phase I/Ib, Open-label, Dose-escalating, Clinical and Pharmacokinetic Study of PM54 Administered Intravenously to Patients With Selected Advanced Solid Tumors.
Brief Title: Clinical Trial of PM54 in Advanced Solid Tumors Patients.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PM54-A-001-22; 2023-508644-22-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-31; First posted 2023-05-03 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PM54 (Experimental): Phase Ia (dose escalation) stage: Patients will receive PM54 i.v. at a starting dose of 0.3 mg/m2.
  Phase Ib (safety run-in) stage: The maximum tolerated dose (MTD) of PM54 previously defined in Phase Ia will be reassessed.
  Phase Ib (expansion) stage: Patients will receive PM54 i.v. at the recommended dose selected after the safety run-in stage.
  Interventions: Drug: PM54

INTERVENTIONS:
Drug: PM54 — PM54 powder for concentrate for solution for infusion (3 mg/vial) is a sterile, preservative-free, lyophilized white to yellowish cake in a single-dose vial for reconstitution prior to intravenous infusion. Each vial contains 3 mg PM54.
  Route of administration: Intravenous infusion

SUMMARY:
The first part of the study (phase Ia - dose escalation) will evaluate the safety and tolerability and identify the dose-limiting toxicities (DLTs) of PM54.

The second part of the study (phase Ib - safety run-in and expansion) will be to reassess the maximum tolerated dose (MTD) defined in the Phase Ia stage in a framework of more extensive premedication, and to evaluate the antitumor activity of PM54 according to the RECIST v.1.1 (or mRECIST v.1.1 in case of MPM) and/or serum markers as appropriate, in patients with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed and dated written informed consent, obtained prior to any specific study procedure.
2. Age ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1.
4. Phase Ia (dose escalation) stage: patients must have:

   1. Pathologically confirmed diagnosis of advanced solid tumors for whom no standard therapy exists:

      * Genitourinary tract tumors: urothelial carcinoma, clear cell renal carcinoma and prostate adenocarcinoma.
      * Cutaneous melanoma.
      * Gastrointestinal: esophageal adenocarcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma, and poorly differentiated (grade 3) gastroenteropancreatic Neuroendocrine Carcinoma (NEC )with Ki67 index >55%.
      * Lung: non-small cell lung cancer (NSCLC) and Small Cell Lung Cancer (SCLC).
      * Gynecological tumors: epithelial ovarian carcinoma (including primary peritoneal disease and/or fallopian tube carcinomas), endometrial adenocarcinoma and carcinoma of cervix.
      * Breast: ductal or lobular.
      * Sarcoma: liposarcoma, leiomyosarcoma, synovial sarcoma and Ewing sarcoma.
      * Deleterious germline BRCA1/2 mutation tumors.
      * Other: MPM, extrapulmonary small cell carcinoma, adrenocortical carcinoma.

      Note: patients with measurable or non-measurable disease according to the Response Evaluation Criteria In Solid Tumors (RECIST) v.1.1 (or mRECIST v.1.1 in case of MPM) are eligible during this stage.
   2. No more than three prior lines of chemotherapy.
5. Phase Ib (safety run-in and expansion) stage: patients must have:

   1. Pathologically confirmed diagnosis of one of the following:

      * Extrapulmonary small cell carcinoma) or poorly differentiated grade 3 gastroenteropancreatic NEC with Ki67 index ≥55%.
      * Cutaneous melanoma.
      * Malignant pleural mesothelioma (MPM).
      * Endometrial adenocarcinoma (Note: carcinosarcomas are not allowed).
      * Synovial sarcoma
   2. Measurable disease according to the RECIST v.1.1 (or mRECIST v.1.1 in case of MPM) and/or evaluable disease byserum markers in case of prostate and ovarian cancer (according to the Prostate-Specific Antigen Working Group Recommendations (PSAWGR) and the Gynecologic Cancer Intergroup (GCIG) specific criteria, respectively).
   3. Progressive disease after last therapy at study entry.
   4. Patients must have received standard treatments:

      * Extrapulomnary small cell carcinoma/ gastroenteropancreatic NEC: no more than two prior lines of chemotherapy.
      * Cutaneous melanoma:

        1. BRAF wild-type (WT) melanoma: at least one prior line of immunotherapy for advanced disease. The patient may have received this therapy in the adjuvant setting. No more than two prior lines of systemic therapy for advanced disease. Note: patients with disease progression during adjuvant therapy or within the first six months after the last dose of adjuvant therapy will be considered as having been treated with one prior line of treatment.
        2. BRAF-mutated melanoma: at least one prior line of target therapy for advanced disease with BRAF inhibitor with or without MEK-inhibitor, and at least one prior line of immunotherapy for advanced disease. The patient may have received any of these therapies in the adjuvant setting. No more than three prior lines of systemic therapy for advanced disease.
      * Malignant pleural mesothelioma (MPM): no more than two prior lines of therapy; one of them should be a platinum containing line. Patients with non-epithelioid MPM should have received a prior immunotherapy line.
      * Endometrial adenocarcinoma: no more than two prior lines of chemotherapy for metastatic disease. In addition, regardless of setting, patients must have received one prior platinum-containing regimen.
      * Synovial sarcoma: at least one but no more than two prior lines of chemotherapy.
6. Recovery to grade ≤1 from drug-related AEs of previous treatments, excluding grade 2 alopecia, according to the NCI-CTCAE v.5.
7. Laboratory values within seven days prior to first infusion:

   1. Absolute Neutrophil Count (ANC) ≥1.5 x 10^9/L, platelet count ≥100 x 10^9/L and hemoglobin ≥9 g/dL (patients may be transfused for anemia as clinically indicated prior to study entry).
   2. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤3.0 x ULN.
   3. Total bilirubin ≤upper limit of normal (ULN) (up to 1.5 x ULN for patients with Gilbert's syndrome).
   4. Creatinine clearance ≥30 mL/min (calculated using the Cockcroft and Gault's formula).
   5. Serum albumin ≥3 g/dL. *
   6. Creatine phosphokinase (CPK) ≤ 2.5 x ULN.
8. Washout periods:

   1. At least three weeks since the last chemotherapy.
   2. At least four weeks since the last monoclonal antibody (MAb)-containing therapy.
   3. At least two weeks since the last biological/investigational single-agent therapy (excluding MAbs) and/or palliative radiotherapy (RT).
   4. In patients with hormone-sensitive breast cancer progressing while on hormone therapy (except for luteinizing hormone-releasing hormone [LHRH] analogues in pre-menopausal women or megestrol acetate), all other hormonal therapies must be stopped at least one week before study treatment start.
   5. Castrate-resistant prostate cancer (CRPC) patients may continue receiving hormone therapy prior to and during study treatment. Note: washout periods will be referred to the day of first cycle administration (Day 1), not to the day of registration.
9. Evidence of non-childbearing status for women of childbearing potential (WOCBP). WOCBP must agree to use a highly effective contraceptive measure during the course of the trial and up to seven months after the last study drug infusion. Fertile male patients with WOCBP partners should use condoms during treatment and for four months following the last study drug infusion.

   * Albumin infusion to increase the blood level in order to fulfill the inclusion criterion is strictly forbidden.

Exclusion Criteria:

For both stages:

1. Concomitant diseases/conditions:

   1. Increased cardiac risk:

      * Uncontrolled arterial hypertension despite optimal management (≥160/100 mmHg).
      * Presence of clinically relevant valvular disease.
      * History of long QT syndrome.
      * Corrected QT interval (QTcF, Fridericia correction) ≥450 ms on screening ECG.
      * History of ischemic heart disease, including myocardial infarction, unstable angina, coronary arteriography or cardiac stress testing with findings consistent with coronary occlusion or infarction ≤6 months prior to study entry.
      * History of heart failure or left ventricular dysfunction (left ventricular ejection fraction [LVEF] ≤50%) by multiple-gated acquisition scan (MUGA) or echocardiography (ECHO).
      * Clinically relevant ECG abnormalities, including any of the following: right bundle branch block with left anterior hemiblock, second (Mobitz II) or third degree atrioventricular block.
      * Symptomatic arrhythmia.
      * Concomitant medication with risk of inducing torsades de pointes, which cannot be discontinued or switched to an alternative drug prior to start PM54 dosing.
      * Use of a cardiac pacemaker.
   2. Active infection requiring systemic treatment.
   3. Known human immunodeficiency virus (HIV) or known chronic active hepatitis. For Hepatitis B, this includes positive tests for both Hepatitis B surface antigen and quantitative Hepatitis B polymerase chain reaction (PCR). For Hepatitis C, this includes positive tests for both Hepatitis C antibody and quantitative Hepatitis C PCR.
   4. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study (e.g., COVID-19).
2. Symptomatic, steroid-requiring, and progressing central nervous system (CNS) disease. Exceptions will be made for patients who have completed radiotherapy at least four weeks prior to inclusion (asymptomatic patients taking steroids in the process of already being tapered within two weeks prior to inclusion).
3. Patients with carcinomatous meningitis.
4. Prior bone marrow or stem cell transplantation.
5. Prior treatment with trabectedin, lurbinectedin, or ecubectedin (PM14).
6. Use of (strong or moderate) inhibitors or strong inducers of CYP3A4 activity within two weeks prior to the first infusion of PM54.
7. Known hypersensitivity to any of the components of the drug product.
8. Limitation of the patient's ability to comply with the treatment or to follow the protocol procedures.
9. Women who are pregnant or breast feeding and fertile patients (men and women) who are not using a highly effective method of contraception (see inclusion criterion No. 9).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1a (dose escalation) and Phase1b (safety run-in): Dose-limiting toxicities (DLTs) | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
Phase 1a (dose escalation) and Phase1b (safety run-in): Treatment-emergent Adverse Events (TEAEs) | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
Phase 1a (dose escalation) and Phase1b (safety run-in): Drug-related Adverse Events (AEs) | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
Phase 1a (dose escalation) and Phase1b (safety run-in): Drug-related deaths | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
Phase 1a (dose escalation) and Phase1b (safety run-in): Serious adverse events (SAEs) | Screening up to end of first cycle of treatment (Cycle 1 is 21 days)
Phase 1a (dose escalation) and Phase1b (safety run-in): Drug-related delays | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
Phase 1a (dose escalation) and Phase1b (safety run-in): Dose reductions | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
Phase 1a (dose escalation) and Phase1b (safety run-in): Treatment discontinuations | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
Phase 1a (dose escalation) and Phase1b (safety run-in): Maximum tolerated dose (MTD) | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
  Lowest dose level explored during dose escalation in which one third (i.e., 33%) or more of evaluable patients develop a DLT in Cycle 1.
Phase 1a (dose escalation) and Phase1b (safety run-in): Recommended dose (RD) | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
  Once the maximum tolerated dose (MTD) is reached, lower dose level will be confirmed as the RD if less than one third (i.e., 33%) of at least nine fully evaluable patients at that dose level develop DLT during Cycle 1.
Phase1b (safety run-in): Determination of RD with more extensive premedication | Day 1 Cycle 1 up to end of first cycle of treatment (Cycle 1 is 21 days)
  A dose level will be confirmed as the RD with more extensive premedication if less than one third (i.e., 33%) of at least nine fully evaluable patients at that dose level develop DLT during Cycle 1.
Phase 1b (expansion): Antitumor activity | Every 6 weeks (± 1 week) in all patients with evaluable disease until Cycle 6. For patients continuing treatment after Cycle 6, assessments performed every 9 weeks (± 1 week) while on treatment, unless otherwise indicated (Up to 48 months)
  Antitumor activity, evaluated according to the RECIST v.1.1 (or mRECIST v.1.1 in case of MPM) and serum markers, as appropriate.

SECONDARY OUTCOMES:
Phase 1b (expansion): Adverse events (AEs) | Screening to end of study (up to approximately 48 months)
  AEs will be graded according to the NCI-CTCAE v.5.
Phase 1b (expansion): Treatment discontinuation | Day 1 up to end of study (up to approximately 48 months)
Phase 1b (expansion): Dose reductions | Day 1 up to end of study (up to approximately 48 months)
Phase 1b (expansion): Treatment delays due to adverse events (AEs) | Day 1 up to end of study (up to approximately 48 months)
Phase 1a (dose escalation) and Phase 1b (safety run-in): QT Assessment | Day 1 of Cycle 1 for all patients participating in the QT assessment, and on Day 1 of Cycle 2 for patients treated during the Phase Ia stage once the MTD has been determined, will be used in this substudy.
  The QT assessment will evaluate the risk of prolongation of the QT interval by PM54.
Phase 1a (dose escalation) and Phase 1b (safety run-in): Maximum Plasma Concentration (Cmax) | Cycle 1 and Cycle 2 during the Phase Ia (dose expansion) stage once the MTD has been determined. Each cycle is 21 days.
Phase 1a (dose escalation) and Phase 1b (safety run-in): Concentration in urine samples | Day 1 of Cycle 1 and Cycle 2 during the Phase Ia (dose expansion) stage once the MTD has been determined. Each Cycle is 21 days.
Phase 1b (safety run-in and dose expansion): Percentage of patients with clinical benefit (overall response rate (ORR) or stable disease (SD) ≥4 months associated with tumor shrinkage) | Day 1 up to end of study (up to approximately 48 months)
Phase 1b (safety run-in and dose expansion): Response rate | Day 1 up to end of study (up to approximately 48 months)
  Response rate defined as percentage of patients with partial response (PR), with complete response (CR), or the sum of both [overall response rate (ORR)].
Phase 1b (safety run-in and dose expansion): Percentage of patients with stable disease (SD) ≥4 months | Day 1 up to end of study (up to approximately 48 months)
Phase 1b (safety run-in and dose expansion): Duration of Response (DoR) | From the date of the first documentation of response to the date of documented progression or death, assessed up to 48 months
Phase 1b (safety run-in and dose expansion): Progression-free Survival (PFS) | From the date of first infusion of study treatment to the date of first documented progression or date of death from any cause, assessed up to 48 months
Phase 1b (safety run-in and dose expansion): Overall survival (OS) | From the date of first infusion of study treatment to the date of death (due to any cause) or last contact (in this case, survival will be censored on the date of last contact), assessed up to 48 months

CONTACTS AND LOCATIONS:
Locations (3):
- South Texas Accelerated Research Therapeutics, San Antonio, Texas, United States
- Institut Jules Bordet, Anderlecht, Belgium
- HM Universitario Sanchinarro, Madrid, M, Spain